CLINICAL TRIAL: NCT06809881
Title: OLFACTION AND BIPOLAR DISODER
Acronym: OLF-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C15-06
Record Dates: First submitted 2017-12-22; First posted 2025-02-05 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2019-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Controls (Other): n= 40 Healthy subjects
  Interventions: Other: olfactory testing, MRI acquisition, clinical assessment
- Patients (Other): n=100 Patients with bipolar disorder
  Interventions: Other: olfactory testing, MRI acquisition, clinical assessment

INTERVENTIONS:
Other: olfactory testing, MRI acquisition, clinical assessment

SUMMARY:
To compare olfactory performance between patients with BD and HC and correlate their performances to neuroimaging data

ELIGIBILITY:
Inclusion Criteria:

* Patients with BD and HC
* Fluent in french
* Having a public health insurance
* Not being on tutorship

Exclusion Criteria:

* Family history of bipolar disorder for controls
* Alcohol dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Olfactive performance | through study completion, an average of 4 years
  Testing of olfactory performance (odor threshold, odor discrimination, odor identification)

CONTACTS AND LOCATIONS:
Locations (1):
- Inserm U 955 Eq 15, Créteil, VAL DE MARNE, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bauer M, Glenn T, Achtyes ED, Alda M, Agaoglu E, Altinbas K, Andreassen OA, Angelopoulos E, Ardau R, Vares EA, Aydin M, Ayhan Y, Baethge C, Bauer R, Baune BT, Balaban C, Becerra-Palars C, Behere AP, Behere PB, Belete H, Belete T, Belizario GO, Bellivier F, Belmaker RH, Benedetti F, Berk M, Bersudsky Y, Bicakci S, Birabwa-Oketcho H, Bjella TD, Brady C, Cabrera J, Cappucciati M, Castro AMP, Chen WL, Cheung EYW, Chiesa S, Crowe M, Cuomo A, Dallaspezia S, Del Zompo M, Desai P, Dodd S, Donix M, Etain B, Fagiolini A, Fellendorf FT, Ferensztajn-Rochowiak E, Fiedorowicz JG, Fountoulakis KN, Frye MA, Geoffroy PA, Gonzalez-Pinto A, Gottlieb JF, Grof P, Haarman BCM, Harima H, Hasse-Sousa M, Henry C, Hoffding L, Houenou J, Imbesi M, Isometsa ET, Ivkovic M, Janno S, Johnsen S, Kapczinski F, Karakatsoulis GN, Kardell M, Kessing LV, Kim SJ, Konig B, Kot TL, Koval M, Kunz M, Lafer B, Landen M, Larsen ER, Lenger M, Lewitzka U, Licht RW, Lopez-Jaramillo C, MacKenzie A, Madsen HO, Madsen SAKA, Mahadevan J, Mahardika A, Manchia M, Marsh W, Martinez-Cengotitabengoa M, Martiny K, Mashima Y, McLoughlin DM, Meesters Y, Melle I, Meza-Urzua F, Ming MY, Monteith S, Moorthy M, Morken G, Mosca E, Mozzhegorov AA, Munoz R, Mythri SV, Nacef F, Nadella RK, Nakanotani T, Nielsen RE, O'Donovan C, Omrani A, Osher Y, Ouali U, Pantovic-Stefanovic M, Pariwatcharakul P, Petite J, Pfennig A, Ruiz YP, Pilhatsch M, Pinna M, Pompili M, Porter R, Quiroz D, Rabelo-da-Ponte FD, Ramesar R, Rasgon N, Ratta-Apha W, Ratzenhofer M, Redahan M, Reddy MS, Reif A, Reininghaus EZ, Richards JG, Ritter P, Rybakowski JK, Sathyaputri L, Scippa AM, Simhandl C, Severus E, Smith D, Smith J, Stackhouse PW Jr, Stein DJ, Stilwell K, Strejilevich S, Su KP, Subramaniam M, Sulaiman AH, Suominen K, Tanra AJ, Tatebayashi Y, Teh WL, Tondo L, Torrent C, Tuinstra D, Uchida T, Vaaler AE, Veeh J, Vieta E, Viswanath B, Yoldi-Negrete M, Yalcinkaya OK, Young AH, Zgueb Y, Whybrow PC. Variations in seasonal solar insolation are associated with a history of suicide attempts in bipolar I disorder. Int J Bipolar Disord. 2021 Sep 1;9(1):26. doi: 10.1186/s40345-021-00231-7. PMID 34467430
- [Background] Favre P, Pauling M, Stout J, Hozer F, Sarrazin S, Abe C, Alda M, Alloza C, Alonso-Lana S, Andreassen OA, Baune BT, Benedetti F, Busatto GF, Canales-Rodriguez EJ, Caseras X, Chaim-Avancini TM, Ching CRK, Dannlowski U, Deppe M, Eyler LT, Fatjo-Vilas M, Foley SF, Grotegerd D, Hajek T, Haukvik UK, Howells FM, Jahanshad N, Kugel H, Lagerberg TV, Lawrie SM, Linke JO, McIntosh A, Melloni EMT, Mitchell PB, Polosan M, Pomarol-Clotet E, Repple J, Roberts G, Roos A, Rosa PGP, Salvador R, Sarro S, Schofield PR, Serpa MH, Sim K, Stein DJ, Sussmann JE, Temmingh HS, Thompson PM, Verdolini N, Vieta E, Wessa M, Whalley HC, Zanetti MV, Leboyer M, Mangin JF, Henry C, Duchesnay E, Houenou J; ENIGMA Bipolar Disorder Working Group. Widespread white matter microstructural abnormalities in bipolar disorder: evidence from mega- and meta-analyses across 3033 individuals. Neuropsychopharmacology. 2019 Dec;44(13):2285-2293. doi: 10.1038/s41386-019-0485-6. Epub 2019 Aug 21. PMID 31434102
- [Background] Sarrazin S, Poupon C, Teillac A, Mangin JF, Polosan M, Favre P, Laidi C, D'Albis MA, Leboyer M, Lledo PM, Henry C, Houenou J. Higher in vivo Cortical Intracellular Volume Fraction Associated with Lithium Therapy in Bipolar Disorder: A Multicenter NODDI Study. Psychother Psychosom. 2019;88(3):171-176. doi: 10.1159/000498854. Epub 2019 Apr 5. PMID 30955011
- [Background] Nunes A, Schnack HG, Ching CRK, Agartz I, Akudjedu TN, Alda M, Alnaes D, Alonso-Lana S, Bauer J, Baune BT, Boen E, Bonnin CDM, Busatto GF, Canales-Rodriguez EJ, Cannon DM, Caseras X, Chaim-Avancini TM, Dannlowski U, Diaz-Zuluaga AM, Dietsche B, Doan NT, Duchesnay E, Elvsashagen T, Emden D, Eyler LT, Fatjo-Vilas M, Favre P, Foley SF, Fullerton JM, Glahn DC, Goikolea JM, Grotegerd D, Hahn T, Henry C, Hibar DP, Houenou J, Howells FM, Jahanshad N, Kaufmann T, Kenney J, Kircher TTJ, Krug A, Lagerberg TV, Lenroot RK, Lopez-Jaramillo C, Machado-Vieira R, Malt UF, McDonald C, Mitchell PB, Mwangi B, Nabulsi L, Opel N, Overs BJ, Pineda-Zapata JA, Pomarol-Clotet E, Redlich R, Roberts G, Rosa PG, Salvador R, Satterthwaite TD, Soares JC, Stein DJ, Temmingh HS, Trappenberg T, Uhlmann A, van Haren NEM, Vieta E, Westlye LT, Wolf DH, Yuksel D, Zanetti MV, Andreassen OA, Thompson PM, Hajek T; ENIGMA Bipolar Disorders Working Group. Using structural MRI to identify bipolar disorders - 13 site machine learning study in 3020 individuals from the ENIGMA Bipolar Disorders Working Group. Mol Psychiatry. 2020 Sep;25(9):2130-2143. doi: 10.1038/s41380-018-0228-9. Epub 2018 Aug 31. PMID 30171211
- [Background] Hibar DP, Westlye LT, Doan NT, Jahanshad N, Cheung JW, Ching CRK, Versace A, Bilderbeck AC, Uhlmann A, Mwangi B, Kramer B, Overs B, Hartberg CB, Abe C, Dima D, Grotegerd D, Sprooten E, Boen E, Jimenez E, Howells FM, Delvecchio G, Temmingh H, Starke J, Almeida JRC, Goikolea JM, Houenou J, Beard LM, Rauer L, Abramovic L, Bonnin M, Ponteduro MF, Keil M, Rive MM, Yao N, Yalin N, Najt P, Rosa PG, Redlich R, Trost S, Hagenaars S, Fears SC, Alonso-Lana S, van Erp TGM, Nickson T, Chaim-Avancini TM, Meier TB, Elvsashagen T, Haukvik UK, Lee WH, Schene AH, Lloyd AJ, Young AH, Nugent A, Dale AM, Pfennig A, McIntosh AM, Lafer B, Baune BT, Ekman CJ, Zarate CA, Bearden CE, Henry C, Simhandl C, McDonald C, Bourne C, Stein DJ, Wolf DH, Cannon DM, Glahn DC, Veltman DJ, Pomarol-Clotet E, Vieta E, Canales-Rodriguez EJ, Nery FG, Duran FLS, Busatto GF, Roberts G, Pearlson GD, Goodwin GM, Kugel H, Whalley HC, Ruhe HG, Soares JC, Fullerton JM, Rybakowski JK, Savitz J, Chaim KT, Fatjo-Vilas M, Soeiro-de-Souza MG, Boks MP, Zanetti MV, Otaduy MCG, Schaufelberger MS, Alda M, Ingvar M, Phillips ML, Kempton MJ, Bauer M, Landen M, Lawrence NS, van Haren NEM, Horn NR, Freimer NB, Gruber O, Schofield PR, Mitchell PB, Kahn RS, Lenroot R, Machado-Vieira R, Ophoff RA, Sarro S, Frangou S, Satterthwaite TD, Hajek T, Dannlowski U, Malt UF, Arolt V, Gattaz WF, Drevets WC, Caseras X, Agartz I, Thompson PM, Andreassen OA. Cortical abnormalities in bipolar disorder: an MRI analysis of 6503 individuals from the ENIGMA Bipolar Disorder Working Group. Mol Psychiatry. 2018 Apr;23(4):932-942. doi: 10.1038/mp.2017.73. Epub 2017 May 2. PMID 28461699